CLINICAL TRIAL: NCT01327222
Title: Intravitreal Bevacizumab for the Treatment of Patients With Low Vision Due to Neovascular Age-related Macular Degeneration
Brief Title: Intravitreal Bevacizumab for Low Vision in Neovascular Age-related Macular Degeneration (AMD)
Acronym: LOW-VISION
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: IRCCS San Raffaele (Other)
Responsible Party: Francesco Bandello, Department of Ophthalmology
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: LOW-VISION
Record Dates: First submitted 2011-03-30; First posted 2011-04-01 (Estimated); Last update posted 2011-04-01 (Estimated); Status verified 2011-01

CONDITIONS: Age Related Macular Degeneration
Keywords: age-related macular degeneration; bevacizumab
MeSH Terms: conditions — Macular Degeneration | interventions — Bevacizumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- bevacizumab (Experimental): three-monthly intravitreal bevacizumab, followed by PRN monthly injection on the basis of the detection of any fluid on the optical coherence tomography
  Interventions: Drug: Bevacizumab
- control (No Intervention): monthly follow-up

INTERVENTIONS:
Drug: Bevacizumab — 1.25 mg intravitreal bevacizumab
  Other Names: avastin
  Arms: bevacizumab

SUMMARY:
The purpose of this study is to compare the effectiveness of intravitreal bevacizumab injection (IVBI) with respect to simple observation in patients with subfoveal choroidal neovascularisation (CNV) secondary to age-related macular degeneration (AMD) presenting at baseline with best corrected visual acuity (BCVA) less than 20/200.

DETAILED DESCRIPTION:
There is no clear indication regarding the treatment of patients with subfoveal choroidal neovascularisation (CNV) secondary to age-related macular degeneration (AMD) presenting at baseline with best corrected visual acuity (BCVA) less than 20/200.

Treatment of eyes with low visual acuity could lead to a waste of resources, without any functional and social improvements.

Aim of the present study is to compare the effectiveness of intravitreal bevacizumab injection (IVBI) with respect to simple observation in

ELIGIBILITY:
Inclusion Criteria:

* age-related macular degeneration
* naïve subfoveal choroidal neovascularization
* best-corrected visual acuity less then 20/200

Exclusion Criteria:

* previous treatments
* any other condition able to limit the visual improvement

Ages: 55 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2011-02; Primary Completion 2011-02 (Actual); Study Completion 2011-02 (Actual)

PRIMARY OUTCOMES:
change in best-corrected visual acuity | 6 months
  change in best-corrected visual acuity at the end of the follow-up

SECONDARY OUTCOMES:
change in central macular thickness | 6 months
  change in central macular thickness on OCT
NEI VFQ-25 scores | 6 months
  change in NEI VFQ-25 scores questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Francesco Bandello, MD, Study Chair — Department of Ophthalmology
Locations (1):
- IRCCS San Raffaele, Milan, MI, Italy

REFERENCES:
- [Background] Arevalo JF, Sanchez JG, Wu L, Berrocal MH, Alezzandrini AA, Restrepo N, Maia M, Farah ME, Brito M, Diaz-Llopis M, Rodriguez FJ, Reategui G, Iturralde-Iraola J, Udaondo-Mirete P; Pan-American Collaborative Retina Study Group. Intravitreal bevacizumab for subfoveal choroidal neovascularization in age-related macular degeneration at twenty-four months: the Pan-American Collaborative Retina Study. Ophthalmology. 2010 Oct;117(10):1974-81, 1981.e1. doi: 10.1016/j.ophtha.2010.01.056. Epub 2010 May 31. PMID 20569989
- [Derived] Parodi MB, Cascavilla M, Papayannis A, Kontadakis DS, Bandello F, Iacono P. Intravitreal bevacizumab in advanced-stage neovascular age-related macular degeneration with visual acuity lower than 20/200. Arch Ophthalmol. 2012 Jul;130(7):934-5. doi: 10.1001/archophthalmol.2011.2617. No abstract available. PMID 22776937